CLINICAL TRIAL: NCT06948214
Title: A Multicenter, 12-Month, Randomized, Double Blind, Placebo-Controlled Phase 3 Efficacy and Safety Study of Daily Oral LUM-201 in Naïve-to-Treatment, Prepubertal Children With Growth Hormone Deficiency (GHD)
Brief Title: Phase 3 Study of LUM-201 in Children With Growth Hormone Deficiency
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Lumos Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LUM-201-10
Record Dates: First submitted 2025-04-21; First posted 2025-04-29 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Growth Hormone Deficiency (GHD)
Keywords: GHD; Pediatric Growth Hormone Deficiency; LUM-201; Growth hormone secretagogue; Height; Catch-up growth; PEM; Oral; Predictive Enrichment Marker; ibutamoren mesylate; OraGrowtH Phase 3 Trial; LUM-201 PEM; GH secretagogue
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- LUM-201 (Experimental)
  Interventions: Drug: LUM-201
- Placebo (Placebo Comparator)
  Interventions: Other: Matched Placebo (Capsules)

INTERVENTIONS:
Drug: LUM-201 — 1.6 mg/kg/day, administered orally once daily
  Arms: LUM-201
Other: Matched Placebo (Capsules) — Administered orally once daily
  Arms: Placebo

SUMMARY:
The OraGrowtH Phase 3 Trial is a multi-national trial. The goals of the trial are to study LUM-201 as a treatment for Pediatric Growth Hormone Deficiency (PGHD) in naive to treatment children and validate the LUM-201 predictive enrichment marker (LUM-201 PEM) strategy to select subjects likely to respond to therapy with daily oral LUM-201.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be naïve to treatment and prepubertal
* Subjects must have a maximal GH response of < 10 ng/mL from 2 prior GH stimulation tests conducted within the preceding 12 months
* Impaired height defined as ≥ 2.0 standard deviations (SDs) below the mean height for chronological age and sex
* Morning or random cortisol level of ≥ 7.0 μg/dL
* ≥ 3.0 years and age ≤ 10.0 years for girls and ≤ 11.0 years for boys
* Baseline height velocity (HV) based on ≥ 6 months of growth assessments < 25th percentile for age and sex
* Bone Age delay of ≥ 12 months compared to the chronological age
* In girls, have genetic testing results to rule out Turner syndrome. If SHOX genetic testing results are available, they need to be negative.
* Have normal thyroid function. Subjects diagnosed with hypothyroidism must have documented successful treatment for at least 3 months prior to Day 1
* Baseline IGF-1 standard deviation score (SDS) ≤ -1.0

Exclusion Criteria:

* Any medical or genetic condition which, in the opinion of the Investigator or Medical Monitor (MM), can be an independent cause of short stature and/or limit the response to exogenous growth factor treatment.
* Arm span to height ratio > 2 SDs below the mean for age and sex
* A medical or genetic condition that, in the opinion of the Investigator and/or MM, adds unwarranted risk to use of LUM-201
* Use of any medication that, in the opinion of the Investigator and/or MM, can independently cause short stature or limit the response to exogenous growth factors
* Current inflammatory diseases requiring systemic corticosteroid treatment for > 2 consecutive weeks within the last 3 months prior to the Screening Visit
* Use of hormone replacement therapy for any hormone deficiency other than thyroid deficiency
* Any ECG at the Screening Visit noted to have a clinically significant abnormality, as confirmed by the MM
* Any subjects suspected of having past or present intracranial tumor growth as confirmed by brain imaging prior to the Screening or Day 1 Visit
* Any subject suspected of having intracranial hypertension (IH) as confirmed by fundoscopy and other assessments
* Any subject with serum alanine transaminase (ALT), aspartate transaminase (AST), or total bilirubin > upper limit of normal (ULN)
* Suspicion of absent pituitary function as evidenced by a maximal stimulated GH ≤ 3.0 ng/mL on any prior standard of care GH stimulation test completed within 12 months
* Body weight ≤ 14.0 kg
* BMI < -2 or > +2 SDs for age and sex based on WHO standards
* Birth weight for gestational age < 3rd percentile based on WHO standards
* Treatment with medications known to be moderate or strong inhibitors or strong inducers of cytochrome P450 (CYP) 3A/4
* History of spinal, cranial, or total body irradiation
* Attention deficit hyperactivity disorder (ADHD) diagnosis

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
AHV after 12 months on LUM-201 compared to placebo | Day 1 to Month 12
  Annualized height velocity (AHV) measured as standing height with stadiometer

OTHER OUTCOMES:
Percentage of subjects selected by PEM strategy who meet target growth | Day 1 to Month 12
  Annualized height velocity (AHV) measured as standing height with stadiometer

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Lumos Pharma Investigational Site, Birmingham, Alabama
  - Lumos Pharma Investigational Site, Sacramento, California
  - Lumos Pharma Investigational Site, Centennial, Colorado
  - Lumos Pharma Investigational Site, Greenwood Village, Colorado
  - Lumos Pharma Investigational Site, Orlando, Florida
  - Lumos Pharma Investigational Site, Tallahassee, Florida
  - Lumos Pharma Investigational Site, New Orleans, Louisiana
  - Lumos Pharma Investigational Site, Las Vegas, Nevada
  - Lumos Pharma Investigational Site, New Brunswick, New Jersey
  - Lumos Pharma Investigational Site, Staten Island, New York
  - Lumos Pharma Investigational Site, Columbia, South Carolina
  - Lumos Pharma Investigational Site, Corpus Christi, Texas
  - Lumos Pharma Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided